CLINICAL TRIAL: NCT07270263
Title: Efficacy and Safety of Reduced-Dose Apixaban and Rivaroxaban Versus Low-Molecular-Weight Heparin in Patients With Hematologic Malignancies: A Prospective Randomized Study
Brief Title: Reduced-Dose Apixaban and Rivaroxaban Versus Low-Molecular-Weight Heparin in Patients With Hematologic Malignancies
Acronym: HEM-DOAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GUM-HEM-DOAC-2025-01
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma; Leukemia; Multiple Myeloma (MM), Lymphoma, Large B-Cell, Diffuse (DLBCL), Lymphoma; Venous Thromboembolic Disease; VTE (Venous Thromboembolism); PE - Pulmonary Embolism; Hematologic Malignacies
Keywords: Apixaban; Rivaroxaban; Low-Molecular-Weight Heparin; Venous Thromboembolism; Cancer-Associated Thrombosis; Hematologic Malignancies; Direct Oral Anticoagulants
MeSH Terms: conditions — Lymphoma; Leukemia; Multiple Myeloma; Venous Thromboembolism; Pulmonary Embolism; Hematologic Neoplasms | interventions — apixaban; Rivaroxaban; Heparin, Low-Molecular-Weight; enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1:1 ratio to receive reduced-dose apixaban, reduced-dose rivaroxaban, or standard low-molecular-weight heparin.
Masking Description: This is an open-label study; no masking will be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- APIXABAN (reduced dose) (Experimental): Participants receive apixaban 2.5 mg orally twice daily for at least 6 months.
  Interventions: Drug: Apixaban
- RIVAROXABAN (reduced dose) (Experimental): Participants receive rivaroxaban 10 mg orally once daily for at least 6 months.
  Interventions: Drug: Rivaroxaban
- Low-Molecular-Weight Heparin (LMWH) (Active Comparator): Participants receive low-molecular-weight heparin, 40 mg subcutaneously once daily for at least 6 months.
  Interventions: Drug: low molecular weight heparin (enoxaparin sodium)

INTERVENTIONS:
Drug: Apixaban — Oral tablet, 2.5 mg twice daily, for at least 6 months.
  Other Names: Eliquis; Poltixa
  Arms: APIXABAN (reduced dose)
Drug: Rivaroxaban — Oral tablet, 10 mg once daily, for at least 6 months.
  Other Names: Xarelto; Mibrex; Zarixa
  Arms: RIVAROXABAN (reduced dose)
Drug: low molecular weight heparin (enoxaparin sodium) — Subcutaneous injection, 40 mg once daily (or equivalent), for at least 6 months.
  Other Names: Clexane; Neoparin
  Arms: Low-Molecular-Weight Heparin (LMWH)

SUMMARY:
This study investigates the efficacy and safety of direct oral anticoagulants (DOACs) in comparison with standard low-molecular-weight heparin (LMWH) for the prevention of venous thromboembolism in patients with hematological malignancies. Eligible participants will be randomized to receive reduced-dose apixaban, reduced-dose rivaroxaban, or standard-dose LMWH. The primary objective is to evaluate the incidence of venous thromboembolism during a 6-month follow-up period. Secondary objectives include assessment of bleeding complications, overall survival, and treatment adherence. The results of this study may provide evidence for safer and more convenient thromboprophylaxis strategies in patients with blood cancers.

DETAILED DESCRIPTION:
Patients with hematologic malignancies are at high risk of developing venous thromboembolism (VTE). Low-molecular-weight heparin (LMWH) is currently the standard of care for thromboprophylaxis in this population; however, daily subcutaneous administration is burdensome and may impair adherence. Direct oral anticoagulants (DOACs), such as apixaban and rivaroxaban, have demonstrated efficacy in the prevention and treatment of VTE in patients with solid tumors, but data in hematologic malignancies are limited.

This study is designed as a prospective, randomized, open-label, parallel-group trial to compare the efficacy and safety of reduced-dose apixaban and rivaroxaban with standard-dose LMWH in patients with hematologic malignancies requiring primary thromboprophylaxis.

Approximately 100 patients will be randomized in a 1:1:1 ratio to receive:

Apixaban 2.5 mg orally twice daily, Rivaroxaban 10 mg orally once daily, or LMWH (enoxaparin 40 mg subcutaneously once daily or equivalent). The primary endpoint is the incidence of symptomatic or objectively confirmed VTE within 6 months of randomization. Secondary endpoints include major and clinically relevant non-major bleeding events (as defined by ISTH), treatment adherence, and overall survival at 6 months.

This study aims to address the unmet clinical need for optimized, patient-friendly thromboprophylaxis in hematologic malignancies and to provide high-quality data that may guide future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Active hematologic malignancy at the time of initiation of systemic therapy, including multiple myeloma, myeloproliferative neoplasm, lymphoma or other hematologic cancer with a Khorana score ≥ 2 points (intermediate or high risk of venous thromboembolism, VTE)
* Use of anticoagulant agents for primary thromboprophylaxis, including direct oral anticoagulants (DOACs) at reduced doses (apixaban 2.5 mg twice daily or rivaroxaban 10 mg once daily) or low-molecular-weight heparin (LMWH) (enoxaparin 40 mg subcutaneously once daily).

Exclusion Criteria:

* Major bleeding within the last month (including gastrointestinal or intracranial bleeding).
* Active major bleeding.
* Hemoglobin concentration < 8 g/dL.
* Thrombocytopenia with platelet count <30 × 10⁹/L.
* ECOG performance status of 3 or 4.
* Expected survival <6 months.
* History of mechanical heart valve or severe mitral stenosis.
* Estimated glomerular filtration rate (eGFR) < 25 mL/min.
* Hepatic impairment (ALT ≥ 3× upper limit of normal or bilirubin ≥ 2× upper limit of normal).
* Acute coronary syndrome or ischemic stroke within the last 6 months.
* Anticipated significant drug-drug interactions between DOACs and anticancer agents.
* Known antiphospholipid syndrome (APS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Venous Thromboembolism (VTE) | 6 months from randomization
  Number of patients who develop symptomatic or incidental venous thromboembolism (deep vein thrombosis or pulmonary embolism) confirmed by objective imaging during the study treatment period.
Incidence of Major Bleeding (ISTH criteria) | 6 months from randomization
  Number of patients experiencing major bleeding as defined by the International Society on Thrombosis and Haemostasis (ISTH).
Incidence of Clinically Relevant Non-Major Bleeding (CRNMB) | 6 months from randomization
  Number of patients experiencing clinically relevant non-major bleeding (CRNMB) according to ISTH definition.

SECONDARY OUTCOMES:
Overall Survival | 6 months
  Proportion of patients alive at 6 months after randomization.
Treatment Discontinuation Due to Adverse Events | 6 months
  Number of patients who discontinued study drug due to adverse events, including bleeding and intolerance.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Haematology & Transplantology, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a non-commercial, single-center academic study with no external data sharing agreements in place.